CLINICAL TRIAL: NCT03378778
Title: The Success and Survival of Teeth and Restoration Following Root Canal Treatment With Varying Degrees of Tooth Structure Loss Restored With CAD CAM Restorations.
Brief Title: Survival of Root Canal Treated Teeth Restored With Ceramic Onlays
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Professor Francesco Mannocci, Professor of Endodontology, King's College London
Other Study IDs: IRAS Project ID: 224248
Record Dates: First submitted 2017-12-05; First posted 2017-12-20 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Dental Pulp Diseases
MeSH Terms: conditions — Dental Pulp Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Less than 33% Tooth Structure remaining: Root canal treatment followed by CAD CAM restoration
  Interventions: Procedure: Root canal treatment
- 33%-50% tooth structure remaining: Root canal treatment followed by CAD CAM restoration
  Interventions: Procedure: Root canal treatment
- 50% -66% tooth structure remaining: Root canal treatment followed by CAD CAM restoration
  Interventions: Procedure: Root canal treatment
- More than 66% tooth structure remaining: Root canal treatment followed by CAD CAM restoration
  Interventions: Procedure: Root canal treatment

INTERVENTIONS:
Procedure: Root canal treatment — Root Canal Treatment followed by Ceramic Onlay restoration

SUMMARY:
Advances in digital dentistry coupled with increased demand for aesthetic restorations have led to developments in CAD CAM( Computer Aided Design and Computer Aided manufacturing)systems for manufacturing tooth restorations. CAD CAM restorations have the added benefit of digital impressions which eliminate the need to take conventional impressions, something patients find difficult to tolerate. CAD CAM restorations are now part of routine dental care. However there are no clinical studies evaluating these restorations on root canal treated teeth

This study aims to compare the success and survival of root canal treated teeth and/or restoration with varying degrees of tooth structure loss restored using CAD CAM restorations.

Null Hypothesis:- The amount of residual coronal dentin has no effect on the survival of root canal treated teeth and/or restoration.

DETAILED DESCRIPTION:
This study will be carried out at KCL Dental Institute at Guy's Hospital and will form part of the routine dental treatment done at the endodontic postgraduate unit. Potential volunteers will be given written information about the process and be given time to consider participation. Once any questions have been answered, fully informed written consent will be obtained if they are interested in taking part. Patients requiring endodontic treatment with varying degrees of tooth structure loss will be detected, diagnosed and treated by endodontic MClinDent postgraduate students at Guy's hospital using suitable clinical techniques. The teeth will then be restored using CAD CAM restorations. Dental periapical radiograph and cone beam computed tomography (CBCT)scans (Morita Accuitomo) will be taken at baseline, 12 months and 24 months. Clinical assessment and radiographical evaluation will be carried out immediately after endodontic treatments have been accomplished and 1 and 2 years post treatment and will be assessed independently by a group of examiners. It is hoped that data analysed from this study will provide a definitive clinical evidence base for the success and survival of endodontically teeth and/or restorations.

ELIGIBILITY:
Inclusion Criteria:

1. Patients either male or female over the age of 18 (who can consent for themselves) in good general health.
2. The selected teeth needed to be in occlusal function with a natural tooth and in interproximal contact with two adjacent natural teeth.
3. Molar or premolar teeth with suspected endodontic problems that require root canal treatment.
4. Teeth should not be mobile and must be restorable.

Exclusion Criteria:

1. Pregnant women, in view of requirements for radiographs (or if they could possibly be pregnant). To be confirmed by the Medical History Questionnaire.
2. Patients younger than 18.
3. Patients unable to give consent.
4. Teeth with probing periodontal depths greater than 5 mm.
5. Non-restorable teeth.
6. Not involving patients from prisons.
7. Not involving patients who cannot read, write or understand English

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Routine patients requiring root canal treatment at Guy's Hospital, London
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Success of root canal treatment | Upto 24 months
  Outcome of root canal treatment assessed using CBCT
Survival of Ceramic Onlays | Upto 24 months
  Survival of ceramic onlays assessed using modified USPHS criteria

SECONDARY OUTCOMES:
Main types of failure of restoration. | Upto 24 months
  Modified USPHS criteria will be used to identify the main types of failure of these restorations.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Mannocci, Principal Investigator — Professor of Endodontology
Locations (1):
- Guy's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data for all primary and secondary outcome measurements will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access requests will be reviewed by an external independent review panel. Requestors will be required to sign a Data Access Agreement

REFERENCES:
- [Background] Al-Nuaimi N, Patel S, Austin RS, Mannocci F. A prospective study assessing the effect of coronal tooth structure loss on the outcome of root canal retreatment. Int Endod J. 2017 Dec;50(12):1143-1157. doi: 10.1111/iej.12760. Epub 2017 Apr 9. PMID 28294354
- [Background] Beier US, Kapferer I, Burtscher D, Giesinger JM, Dumfahrt H. Clinical performance of all-ceramic inlay and onlay restorations in posterior teeth. Int J Prosthodont. 2012 Jul-Aug;25(4):395-402. PMID 22720292

DOCUMENTS (3):
  • Study Protocol (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/78/NCT03378778/Prot_000.pdf
  • Informed Consent Form (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/78/NCT03378778/ICF_001.pdf
  • Statistical Analysis Plan (2017-12-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT03378778/SAP_002.pdf